CLINICAL TRIAL: NCT02358356
Title: Capecitabine ON Temozolomide Radionuclide Therapy Octreotate Lutetium-177 NeuroEndocrine Tumours Study
Acronym: CONTROL NETS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Australasian Gastro-Intestinal Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTC0120 / AG0114NET
Record Dates: First submitted 2014-11-04; First posted 2015-02-09 (Estimated); Last update posted 2022-07-05 (Actual); Status verified 2017-11

CONDITIONS: Midgut Neuroendocrine Tumours; Pancreatic Neuroendocrine Tumours
Keywords: midgut; pancreatic; neuroendocrine; advanced; unresectable low; intermediate grade; mNETs; pNETs
MeSH Terms: conditions — Neuroectodermal Tumors, Primitive | interventions — Capecitabine; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PRRT (Active Comparator): 7.8GBq 177Lu Octreotate (Lutate) given intravenously (IV) on day 1 every 8 weeks for 4 cycles.
  Interventions: Drug: octreotate
- CAPTEM (Active Comparator): Oral capecitabine 750mg/m2 b.i.d. days 1-14 and temozolomide 75mg/m2 b.i.d. days 10-14 every 28 day cycle, up to 8 cycles.
  Interventions: Drug: Capecitabine; Drug: Temozolomide
- PRRT/CAPTEM (Experimental): 7.8GBq 177Lu Octreotate (Lutate) given intravenously (IV) on day 10 every 8 weeks for 4 cycles, with concurrent oral capecitabine 750mg/m2 b.i.d. days 1-14 and temozolomide 75mg/m2 b.i.d. days 10-14 up to 4 cycles.
  Interventions: Drug: octreotate; Drug: Capecitabine; Drug: Temozolomide

INTERVENTIONS:
Drug: octreotate — 7.8GBq 177Lu Octreotate (Lutate) given intravenously (IV)
  Other Names: lutate
  Arms: PRRT; PRRT/CAPTEM
Drug: Capecitabine — oral capecitabine 750mg/m2 b.i.d.
  Other Names: Xeloda
  Arms: CAPTEM; PRRT/CAPTEM
Drug: Temozolomide — temozolomide 75mg/m2 b.i.d.
  Arms: CAPTEM; PRRT/CAPTEM

SUMMARY:
Two parallel phase II randomized open label trials of Lutetium-177 Octreotate (177Lu-Octreotate) peptide receptor radionuclide therapy (PRRT) and capecitabine (CAP)/temozolomide (TEM) chemotherapy (chemo): (i) versus CAPTEM alone in the treatment of low to intermediate grade pancreatic neuroendocrine tumours (pNETs); (ii) versus PRRT alone in the treatment of low to intermediate grade mid gut neuroendocrine tumours (mNETs).

DETAILED DESCRIPTION:
PROTOCOL SYNOPSIS

Background

Neuroendocrine tumours (NETs) are a heterogeneous group of malignancies that can arise at any site in the gastrointestinal tract, that are known by their ability to over express somatostatin receptors. Originally called carcinoid tumours, these tumours are rising in incidence. In patients with incurable disease, several systemic options have demonstrated activity but few have been compared in prospective, randomised controlled trials (RCTs). 177Lu-Octreotate peptide receptor radionuclide therapy (PRRT) and CAPTEM have shown promising activity in initial single arm trials. Prospective RCTs are needed to build on these early trials to determine the optimal role of these therapies in clinical practice.

CONTROL NETs is a parallel group phase II randomised open label trial of Lutetium-177 Octreotate (177Lu-Octreotate (Lutate)) peptide receptor radionuclide therapy (PRRT) and capecitabine (CAP)/temozolomide (TEM) chemotherapy (chemotherapy): (i) versus CAPTEM alone in the treatment of low to intermediate grade pancreatic neuroendocrine tumours (pNETs); (ii) versus PRRT alone in the treatment of low to intermediate grade midgut neuroendocrine tumours (mNETs).

General aim

i) To determine the relative activity of CAPTEM/PRRT in biopsy-proven, low to intermediate grade, unresectable, metastatic 68Ga-octreotate PET-avid NETs in the following parallel phase II studies: Group A: pNETs and Group B: mNETs.

ii) To inform future comparative phase III RCTs to determine the optimal therapies in pNETs and mNETs.

Design

Two parallel non-comparative group randomised, controlled, multi-centre phase II, 2 arm open-label controlled trials with 2:1 allocation (experimental : control)

1. Study A: pNETs: PRRT/CAPTEM vs. CAPTEM (control)
2. Study B: mNETs: PRRT/CAPTEM vs. PRRT (control)

Randomisation will be performed using the method of minimisation.

Patients will be stratified by:

* Previous systemic therapy regimens (0,1 v 2)
* WHO tumour grade: Low Grade - G1 (Ki67<3% (mitotic count <2)) vs. Intermediate Grade - G2 (Ki67 3-20% (mitotic count 2-20))
* visceral only vs. visceral with bone metastases
* Treating institution

Population

The target population for this study is consenting adult patients with advanced, unresectable low or intermediate grade (Ki-67<20%) midgut neuroendocrine tumours (mNETs) or pancreatic neuroendocrine tumours (pNETs ), who have received ≤ 2 prior systemic therapies for advanced unresectable disease (including long acting somatostatin analogues).

Assessments

* Patients will be assessed at each treatment cycle for toxicity
* CT including a 3 phase contrast CT of the liver will be undertaken at baseline, then every 2 months (pNET) or every 4 months (pNET) until radiologic progression by RECIST v1.1.
* 68Ga-DOTATATE PET CT Scan will be undertaken at baseline, then every 4 months until radiologic progression by RECIST v1.1.
* 18F-FDG PET Scan may be performed at the discretion of treating clinician at baseline, then every 2 months until radiologic progression by RECIST v1.1) for G2 NETS.
* 24-h whole-body planar gamma imaging will be undertaken on the day after administration of PRRT (every 2 months).
* Serum biomarkers will be undertaken every 4 months until disease progression.
* Quality of life assessments will be undertaken at every 2 months until disease progression using QLC C30 and QLQ-GINET21.
* Health utilities will be evaluated with EQ-5D-5L every 2 months until completion of study follow up.

Statistical considerations

Both studies are based on a Simon's two-stage design and are randomised using a 2:1 randomisation (Experimental: Control). A mix of approximately 30% G1 patients and 70% G2 patients is expected.

Study A, pNETs (n=90) will have 80% power with 95% confidence interval to exclude a 12 months PFS of 60% in favour of a more interesting rate of 77% in the experimental arm.

For Study B, mNETs (n=75), the PFS at 24 months in the control arm is expected to be 52%. Thus study B will have 80% power with 95% confidence interval to demonstrate a PFS rate at 24 months of 70% in experimental arm, a result that would warrant further investigation.

A total sample size of 165 patients for the two studies will be accrued over 2 years.

Patients will be followed up for a minimum of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years old with histologically proven, moderate to well-differentiated G1/2 pancreatic or midgut NETs with Ki-67 < 20%;
* The presence of somatostatin receptor avidity suitable for PRRT demonstrated on 68Ga-octreotate PET scan;
* Progressive advanced/metastatic disease that has progressed during or after ≤ 2 prior systemic therapies;
* Unresectable disease, determined by an appropriately specialized surgeon or deemed not suitable for liver directed therapies where liver is the only site of disease;
* ECOG performance status 0-2;
* Ability to swallow oral medication;
* Adequate renal function (measured creatinine clearance > 50 ml/min by DTPA or 51CR-EDTA), bone marrow function (Hb > 9 g/d/L, ANC > 1.5 x109L, and platelets > 100 x 10/L);
* Adequate liver function (serum total bilirubin ≤ 1.5 x ULN, and Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), Alkaline phosphatase (ALP) ≤ 2.5 x ULN (≤ 5 x ULN for patients with liver metastases)). INR ≤ 1.5 (or on a stable dose of LMW heparin for >2 weeks at time of enrolment .);
* Life expectancy of at least 9 months;
* Study treatment both planned and able to start within 28 days of randomisation; )
* Willing and able to comply with all study requirements, including treatment, timing and/or nature of required assessments;
* Signed, written informed consent.

Exclusion Criteria:

* Primary NETs other than small bowel (midgut) or pancreatic NETs;
* Cytotoxic chemotherapy, targeted therapy, or biotherapy within the last four weeks;
* Prior intrahepatic 90Y microspheres, such as SIR-Spheres in the past six months;
* Prior Peptide Receptor Radionuclide Therapy;
* Major surgery/surgical therapy for any cause within one month;
* Surgical therapy of loco-regional metastases within the last three months prior to randomisation;
* Uncontrolled metastatic disease to the central nervous system. To be eligible, CNS metastases should have been treated with surgery and/or radiotherapy and the patient should have been receiving a stable dose of steroids for at least 2 weeks prior to randomisation, with no deterioration in neurological symptoms during this time;
* Poorly controlled concurrent medical illness. E.g. unstable diabetes (Note: optimal glycaemic control should be achieved before starting trial therapy); Symptomatic NYHA class III or IV congestive cardiac failure, myocardial infarction within 6 months of start of the study, serious uncontrolled cardiac arrhythmia, unstable angina, or any other clinically significant cardiac disease;
* History of other malignancies within 5 years except where treated with curative intent AND with no current evidence of disease AND considered not to be at risk of future recurrence Patients with a past history of adequately treated carcinoma-in-situ, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or superficial transitional cell carcinoma of the bladder are eligible;
* Any uncontrolled known active infection, including chronic active hepatitis B, hepatitis C, or HIV. Testing for these is not mandatory unless clinically indicated. Participants with known Hepatitis B/C infection will be allowed to participate providing evidence of viral suppression has been documented and the patient remains on appropriate anti-viral therapy;
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of capecitabine/temozolomide (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or substantial small bowel resection);
* Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule, including alcohol dependence or drug abuse;
* Pregnancy, lactation, or inadequate contraception. Women must be post-menopausal, infertile, or use a reliable means of contraception. Women of childbearing potential must have a negative pregnancy test done within 7 days prior to registration. Men must have been surgically sterilised or use a (double if required) barrier method of contraception .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-11; Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 12 months for pNETs and 24 months for mNets
  To determine the rate of progression free survival (PFS) at 12 months in pNETs (Group A), and at 24 months in mNETs (Group B). (PFS defined from time of randomisation to disease progression as defined by RECIST criteria version 1.1).

SECONDARY OUTCOMES:
Objective tumour response rate (partial or complete response) as per RECIST v1.1 criteria | 12 months or 24 months as appropriate
  To determine objective tumour response rate (OTRR) (partial or complete response (PR/CR)).
Overall survival (death from any cause) | 12 months or 24 months as appropriate
  To determine overall survival (OS) (death from any cause).
Safety (rates of adverse events worst grade according to NCI CTCAE v4.0) | 12 months or 24 months as appropriate
  To determine safety (rates of adverse events).
Quality of life (QOL scores determined at beginning, during treatment and until disease progression) | 12 months or 24 months as appropriate
  To determine Quality of Life (QoL) (QoL scores from EORTC QLQ C30 and QLQ-GINET21 questionnaires)
Resource utilisation (use of healthcare resources) and cost-effectiveness (Health utility score determined at beginning, during treatment and until end of follow up, correlated with MBS & PBS data) | 12 months or 24 months as appropriate
  To determine resource utilization (costs associated with treatment regimen, MBS and PBS data, and health utilities scores from EQ-5D-5L).
Clinical Benefit | 12 months or 24 months as appropriate
  To evaluate the proportion of patients who have experienced a clinical benefit of the regimen(s). (Clinical Benefit is defined as the proportion of patients who experience complete or partial response (using RECIST v1.1) or stable disease at 12 months or 24 months as appropriate).

OTHER OUTCOMES:
biomarkers CgA, Ki-67 and tumour MGMT expression with survival, response and safety. | 12 months or 24 months as appropriate
  To correlate circulating & tissue biomarkers with clinical study endpoints (relating to survival, response and safety), including but not limited to CgA, Ki-67 & tumour MGMT expression.
Other measures of response such as 68Ga-DOTATATE, SUVmax, tumour update and other measures of response of a biochemical measure such as tumour markers, chomogranin A and patient reported outcomes. | 12 months or 24 months as appropriate
  Explore correlation between other measures of response relevant to this disease, eg 68Ga-DOTATATE, SUVmax tumour uptake, and other measures of response of a biochemical measure, eg. tumour markers, chromogranin A, and patient reported outcomes QOL undertaken in order to identify how progressive symptoms or biochemical response relates to conventional measures of response using structural and/or functional imaging. A formal statistical analysis plan will be formulated prior to final data analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Nick Pavlakis, Associate Professor, Study Chair — Royal North Shore Hospital
Locations (4):
- Australia (4):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia